CLINICAL TRIAL: NCT01247857
Title: Double Blind Randomized Phase III Controlled Trial Comparing the Effect of Preoperative and Postoperative Nebulization of Ropivacaine on Pain Control After Laparoscopic Cholecystectomy
Brief Title: Local Anesthetic Nebulization for Pain Control After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Collaborators: Hôpital de Hautepierre (Other)
Responsible Party: Pablo M Ingelmo, MD, First Service of anesthesia and intensive care. San Gerardo Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR HSG 02-2008
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2008-03

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; Nebulization; Ropivacaine
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Preoperative Nebulization (Active Comparator): Nebulization of 30 mg of Ropivacaine in the peritoneal cavity before surgery
  Interventions: Drug: Ropivacaine 30 mg
- Postoperative Nebulization (Active Comparator): Nebulization of 30 mg of Ropivacaine in the peritoneal cavity after surgery
  Interventions: Drug: Ropivacaine 30 mg
- Control (Placebo Comparator): Nebulization of normal saline 3 ml before and after surgery
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine 30 mg — Intraperitoneal nebulization of ropivacaine 1% 3 ml (30 mg) before surgery and intraperitoneal nebulization of normal saline 3 ml after surgery.
  Nebulization was performed over 5-10 minutes using the Aeroneb Pro® device through the umbilical port during the insertion of the other ports, while postoperative nebulization was performed before the withdrawal of the ports.
  Arms: Preoperative Nebulization
Drug: Ropivacaine 30 mg — intraperitoneal Nebulization of normal saline 3 ml before surgery and intraperitoneal nebulization of ropivacaine 1% 3 ml (30 mg) after surgery.
  Nebulization was performed over 5-10 minutes using the Aeroneb Pro® device through the umbilical port during the insertion of the other ports, while postoperative nebulization was performed before the withdrawal of the ports.
  Arms: Postoperative Nebulization
Drug: Saline — Intraperitoneal nebulization of normal saline 3 ml before and after surgery. Nebulization was performed over 5-10 minutes using the Aeroneb Pro® device through the umbilical port during the insertion of the other ports, while postoperative nebulization was performed before the withdrawal of the ports.
  Arms: Control

SUMMARY:
Intraperitoneal nebulization of local anesthetic is a novel approach to pain management after laparoscopy. Preoperative compared with postoperative administration of analgesia remains controversial. This randomized, double blind, placebo-controlled trial compared the analgesic efficacy of preoperative with postoperative peritoneal ropivacaine nebulization in patients undergoing elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Previous studies evaluating intraperitoneal local anesthetic administration for pain relief after laparoscopic surgery have suggested that the timing of local anesthetic administration may be critical in the success of the technique. A meta-analysis of randomized trials of intraperitoneal local anesthetic instillation in patients undergoing laparoscopic surgery found that local anesthetic instilled before surgical dissection provided superior pain relief compared to instillation at the end of surgery. Intraperitoneal nebulization of local anesthetic is a novel approach to pain management after laparoscopic surgery. Recently, Alkhamesi et al reported that bupivacaine nebulization performed at the end of laparoscopic cholecystectomy significantly reduced postoperative pain. However, clinical benefits of preoperative administration of analgesia, compared with postoperative administration, remains controversial.

The investigators hypothesized that pain relief after preoperative and postoperative ropivacaine nebulization would be similar but better than placebo.

ELIGIBILITY:
Inclusion Criteria:

* ASA Score I-III
* Scheduled for laparoscopic cholecystectomy
* Free from pain in preoperative period
* Not using analgesic drugs before surgery
* Without cognitive impairment or mental retardation
* Written informed consent

Exclusion Criteria:

* Emergency/urgency surgery
* Postoperative admission in an intensive care unit
* Cognitive impairment or mental retardation
* Progressive degenerative diseases of the CNS
* Seizures or chronic therapy with antiepileptic drugs
* Severe hepatic or renal impairment
* Pregnancy or lactation
* Allergy to one of the specific drugs under study
* Acute infection or inflammatory chronic disease
* Alcohol or drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 48 hours
  Postoperative pain will be assessed by numeric ranking scale (NRS 0 to 10 points) at rest (static NRS) and after a deep inspiration or cough (dynamic NRS). The proportion of patients with adequate pain control after surgery (dynamic NRS < 3) will also be assessed.

SECONDARY OUTCOMES:
Time of unassisted walking | Up to 48 hours
  Unassisted walking time is defined as the time in hours between PACU discharge and when the patient is able to walk out of his room and back to bed without any assistance.
Morphine consumption (mg) | Up to 48 hours
  The total dose of morphine at every evaluation after awakening will be quantified using the PACU clinical chart and/or PCA infusers memory display
Hospital morbidity | Up to 48 hours
  All complications or adverse effects associated or possibly associated with the interventions under study, surgery or anesthesia will be quantified using the anesthesia charts, surgical charts, surgical database.
Time to hospital discharge | 48 hours
  We define hospital stay as the elapsed time between surgery and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Ingelmo, MD, Principal Investigator — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Result] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Result] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034
- [Result] Schlotterbeck H, Schaeffer R, Dow WA, Diemunsch P. Cold nebulization used to prevent heat loss during laparoscopic surgery: an experimental study in pigs. Surg Endosc. 2008 Dec;22(12):2616-20. doi: 10.1007/s00464-008-9841-z. Epub 2008 Mar 18. PMID 18347861